CLINICAL TRIAL: NCT05410938
Title: Triweekly Chemotherapy With Bevacizumab Versus Intraperitoneal Chemotherapy as Frontline Therapy in Advanced Ovarian Cancer
Brief Title: Intraperitoneal Chemotherapy Versus Triweekly Chemotherapy
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief of Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 111113-E
Record Dates: First submitted 2022-06-06; First posted 2022-06-08 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Intraperitoneal Chemotherapy, Bevacizumab, Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intraperitoneal group: The intraperitoneal regimen was given as 135 mg/m2 intravenous paclitaxel over a 3 or 24 hours period on day 1, followed by 75-100 mg/m2 intraperitoneal cisplatin on day 2 and 60 mg/m2 intraperitoneal paclitaxel on day 8. For women with significantly impaired renal function (i.e., estimated glomerular filtration rate<50 mL/min/1.73 m2), carboplatin (area under the curve [AUC]=6) was used instead of cisplatin.
  Interventions: Drug: Chemotherapy
- Triweekly group: The triweekly intravenous chemotherapy regimen was given as 175 mg/m2 paclitaxel and carboplatin at a dose calculated to produce an AUC of 6 mg/mL/min on day 1. Bevacizumab was given at a dose of 7.5mg/kg intravenously on day 2 since cycle 2. The treatments were repeated every 3 weeks for 6 cycles. Those women without achievement of complete response after 6 cycles of chemotherapy might be treated with an additional 1-2 cycles of chemotherapy. Bevacizumab was continued for 12 additional cycles or until disease progression, death, unacceptable toxic effects, or patient voluntary withdrawal [5].
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Triweekly chemotherapy with bevacizumab versus intraperitoneal chemotherapy without bevacizumab

SUMMARY:
The combination of paclitaxel and carboplatin is the standard first-line chemotherapy for ovarian cancer as recommended by the NCCN Guidelines for Epithelial Ovarian Cancer, and is conventionally given via intravenous route every three weeks. The addition of target therapy (bevacizumab) has shown to improve progression free survival but not overall survival. Several trials have also demonstrated a clinically significant survival advantage associated with intraperitoneal chemotherapy compared to intravenous chemotherapy, and the best outcomes are consistently seen for patients who have no residual disease. This study aims to compare triweekly chemotherapy with bevacizumab versus intraperitoneal chemotherapy in patients with advanced stage ovarian cancer.

ELIGIBILITY:
Inclusion Criteria:

* women aged 20 and above with FIGO stage II-IV advanced ovarian, fallopian tube or primary peritoneal cancer who received debulking surgery, followed by either triweekly intravenous chemotherapy with bevacizumab or intraperitoneal chemotherapy; women who received neoadjuvant chemotherapy followed by interval debulking surgery were also eligible for participation. Intraperitoneal chemotherapy was defined as having one or more cycles of an intraperitoneal regimen administered.

Exclusion Criteria:

* women who quit half-way or received chemotherapy at other site

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — women aged 20 and above with FIGO stage II-IV advanced ovarian, fallopian tube or primary peritoneal cancer
Study Population: women aged 20 and above with FIGO stage II-IV advanced ovarian, fallopian tube or primary peritoneal cancer
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival | the time interval from the date of surgery or neoadjuvant chemotherapy to clinically defined recurrence, disease progression, or the last follow-up

SECONDARY OUTCOMES:
Overall survival | the time interval from the date of surgery or neoadjuvant chemotherapy to the date of death from any cause or the last follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No